CLINICAL TRIAL: NCT06360133
Title: A Phase 3, Randomized, Double-Masked, Vehicle-controlled, Multi-center Study Evaluating the Safety and Efficacy of 5% VVN001 in Chinese Subjects With Dry Eye Disease
Brief Title: Study of 5% VVN001 Ophthalmic Solution in Dry Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN001-CCS-301
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VVN001 (Experimental): VVN001 Ophthalmic Solution, 5%
  Interventions: Drug: VVN001 Ophthalmic Solution, 5%
- Vehicle (Placebo Comparator): VVN001 Ophthalmic Solution, Vehicle
  Interventions: Drug: VVN001 Ophthalmic Solution, Vehicle

INTERVENTIONS:
Drug: VVN001 Ophthalmic Solution, 5% — VVN001 Ophthalmic Solution, 5%
  Arms: VVN001
Drug: VVN001 Ophthalmic Solution, Vehicle — VVN001 Ophthalmic Solution, Vehicle
  Arms: Vehicle

SUMMARY:
This is a Phase 3, randomized, double-Masked, vehicle-controlled, multi-center study designed to evaluate the safety and efficacy of 5% VVN001 Ophthalmic Solution versus vehicle in Chinese subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent prior to any study-related procedures.
* Are between 30 and 80 years of age.
* Have a history of dry eye disease in both eyes.
* Have been using artificial tears within 30 days of the screening visit
* Have an Eye dryness score ≥50 (0-100 point VAS)
* Have ongoing dry eye disease in the same eye or both eyes, as defined by all of the following criteria in the study eye and the same eye at Visit 1 and Visit 2: 1) total CFS (tCFS) score ≥6; 2) any subregion CS score ≥2.5; 3) Schirmer score (without anesthesia) ≥1 and ≤7 mm/5 min.
* Have a BCVA in the study eye of ≥4.3 (Standard for Logarithmic Visual Acuity Charts, 5-mark record).

Exclusion Criteria:

* Have a known hypersensitivity or contraindication to the IP or components of IP.
* Have history of uncontrolled glaucoma, IOP over 21 mmHg in either eye at the screening visit or are being treated with eye drops for glaucoma in the study eye. Or the subject has had laser or surgery for glaucoma in the study eye within 90 days of the study.
* Woman of childbearing potential (WOCP) who are pregnant, lactating, or preparing for pregnant.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | Day 84
  Mean Change from baseline (Visit 2) to Day84 (Visit 6) in total corneal fluorescein staining (tCFS) using modified NEI/Industry Workshop (0-4 scale, using 0.5 unit increments).

SECONDARY OUTCOMES:
Eye Dryness | Day 84
  Mean Change from baseline (Visit 2) to Day 84 (Visit 6) in the individual symptom of eye dryness (0~100 VAS scale).

CONTACTS AND LOCATIONS:
Overall Officials: Xinghuai Sun, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & Ent Hospital of Fudan University, Shanghai, Shanghai Municipality, China